CLINICAL TRIAL: NCT04737824
Title: Immediate and Long-term Effects of an Adaptation of the "Balloon-blowing Exercise" on the Thoracoabdominal Movement in Healthy Students - a Randomized Controlled Trial
Brief Title: Immediate and Long-term Effects of an Adaptation of the "Balloon-blowing Exercise"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, António Manuel Soares Mesquita Montes, Principal Investigator, Escola Superior de Tecnologia da Saúde do Porto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESS-Balloon
Record Dates: First submitted 2021-01-30; First posted 2021-02-04 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental group A (Experimental): Participants executed two sets of twelve repetitions of an adaptation of the "balloon-blowing" exercise.
  Interventions: Procedure: An adaptation of the "balloon-blowing" exercise
- Control group A (No Intervention): No intervention was applied.
- Experimental group B (Experimental): Participants executed two sets of twelve repetitions of an adaptation of the "balloon-blowing" exercise for seven weeks, three times a week, at home.
  Interventions: Procedure: An adaptation of the "balloon-blowing" exercise for seven weeks, three times a week, at home
- Control group B (No Intervention): No intervention was applied.

INTERVENTIONS:
Procedure: An adaptation of the "balloon-blowing" exercise — The participants were positioned in supine, on a semi-rigid surface, with the upper limbs placed above the level of the head, at rest. Their feet were also placed at a resting position on a wall and with their hips and knees at 90o of flexion. The cervical was placed in a neutral position and the pelvis was maintained in a posterior pelvic tilt, both structures corrected by the researcher. The participants were asked to contract the adductors, maintaining a bilateral and symmetric pressure between 10 and 15 mmHg on two sphygmomanometers placed between the knees. Also, an isometric contraction of the hamstrings and gluteus was requested. A Threshold®, with a minimum resistance of 5 cmH2O, and they were instructed to close their lips around the mouthpiece, to avoid air leaks. To start the exercise, it was transmitted to the participants to make a maximum inspiration through the nose, for two seconds. Subsequently, a maximum exhalation throughout the threshold was made for three seconds.
  Other Names: Motor control exercise A
  Arms: Experimental group A
Procedure: An adaptation of the "balloon-blowing" exercise for seven weeks, three times a week, at home — The participants were positioned in supine, on a semi-rigid surface, with the upper limbs placed above the level of the head, at rest. Their feet were also placed at a resting position on a wall and with their hips and knees at 90o of flexion. The cervical was placed in a neutral position and the pelvis was maintained in a posterior pelvic tilt, both structures corrected by the researcher. The participants were asked to contract the adductors, maintaining a bilateral and symmetric pressure between 10 and 15 mmHg on two sphygmomanometers placed between the knees. Also, an isometric contraction of the hamstrings and gluteus was requested. A Threshold®, with a minimum resistance of 5 cmH2O, and they were instructed to close their lips around the mouthpiece, to avoid air leaks. To start the exercise, it was transmitted to the participants to make a maximum inspiration through the nose, for two seconds. Subsequently, a maximum exhalation throughout the threshold was made for three seconds.
  Other Names: Motor control exercise B
  Arms: Experimental group B

SUMMARY:
Despite the literature evidence that the "balloon-blowing exercise" improves the pulmonary function as a long-term effect, this exercise has not yet been studied or tested experimentally, meaning that there are no specific and measurable results that attest the improvement on thoracoabdominal movement.

ELIGIBILITY:
The target population consisted of healthy physiotherapy students from School of Health - Polytechnic of Porto, who volunteered to participate in study.

Inclusion criteria:

- In the Experimental Group B were admitted individuals that, through the analysis of the training record sheet, had executed 2⁄3 of the programmed sessions.

Exclusion criteria:

* Individuals that had participated in aerobic physical activities of moderate (i.e., at least 30 minutes on five days per week) or vigorous intensity (i.e., at least 20 minutes on three days per week) for more than one year;
* Chronic nonspecific lumbopelvic pain (i.e., recurrent episodes of lumbopelvic pain for a period exceeding three months);
* Flu symptoms or respiratory infection up to one week before data collection;
* History of recent ribs fracture and pain in the last three months;
* Pulmonary or rib cage previous pathologies;
* Length discrepancy of the lower limbs or other postural asymmetries;
* History of spinal, gynaecological, or abdominal surgery in the previous year;
* Recurrent muscle/joint pain and history of musculoskeletal injury in the last three months;
* Smoking and/or drinking habits.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Anterior-to-posterior movement of the upper rib cage | Immediate after procedure
  Thoracoabdominal movement was measure through "Qualisys motion capture system".
Anterior-to-posterior movement of the lower rib cage | Immediate after procedure
  Thoracoabdominal movement was measure through "Qualisys motion capture system".
Anterior-to-posterior abdominal movement | Immediate after procedure
  Thoracoabdominal movement was measure through "Qualisys motion capture system".
Medial-to-lateral movement of the upper rib cage | Immediate after procedure
  Thoracoabdominal movement was measure through "Qualisys motion capture system".
Medial-to-lateral movement of the lower rib cage | Immediate after procedure
  Thoracoabdominal movement was measure through "Qualisys motion capture system".
Anterior-to-posterior movement of the upper rib cage | Seven weeks
  Thoracoabdominal movement was measure through "Qualisys motion capture system".
Anterior-to-posterior movement of the lower rib cage | Seven weeks
  Thoracoabdominal movement was measure through "Qualisys motion capture system".
Anterior-to-posterior abdominal movement | Seven weeks
  Thoracoabdominal movement was measure through "Qualisys motion capture system".
Medial-to-lateral movement of the upper rib cage | Seven weeks
  Thoracoabdominal movement was measure through "Qualisys motion capture system".
Medial-to-lateral movement of the lower rib cage | Seven weeks
  Thoracoabdominal movement was measure through "Qualisys motion capture system".

CONTACTS AND LOCATIONS:
Locations (1):
- Escola Superior de Saúde - Instituto Politécnico do Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Boyle KL, Olinick J, Lewis C. The value of blowing up a balloon. N Am J Sports Phys Ther. 2010 Sep;5(3):179-88. PMID 21589673
- [Background] De Troyer A. Respiratory effect of the lower rib displacement produced by the diaphragm. J Appl Physiol (1985). 2012 Feb;112(4):529-34. doi: 10.1152/japplphysiol.01067.2011. Epub 2011 Dec 1. PMID 22134697
- [Background] Key J. 'The core': understanding it, and retraining its dysfunction. J Bodyw Mov Ther. 2013 Oct;17(4):541-59. doi: 10.1016/j.jbmt.2013.03.012. Epub 2013 Jun 28. PMID 24139017